CLINICAL TRIAL: NCT04596384
Title: Comparative Effectiveness Trial of Perioperative Telemonitoring for Functional Recovery and Symptoms
Brief Title: Home Base Telemonitoring in Gastrointestinal, Genitourinary, or Gynecologic Cancer Patients Undergoing Abdominal Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20370; NCI-2020-07889 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20370 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Digestive System Carcinoma; Genitourinary System Carcinoma; Malignant Female Reproductive System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (telemonitoring program, actigraph, TapCloud) (Experimental): Before surgery, patients complete a functional and nutritional assessment. The home environment of patients will also be assessed. Based on findings, patients undergo personalized prehabilitation. Patients also wear an actigraph throughout the study to measure and record daily steps taken and sedentary time. Patients use the TapCloud app on a smart device (phone, tablet) or home computer to collect, track, and report their symptoms. Based on patient input in the TapCloud app, a real-time alert is sent to an RN when predetermined thresholds are met. RNs then contact the patient via the TapCloud app and further phone calls if necessary. Patients, caregivers and surgeons may also participate in a focus group in-person, via telephone, or videoconferencing.
  Interventions: Procedure: Functional Assessment; Other: Medical Device Usage and Evaluation; Procedure: Nutritional Assessment; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: TapCloud
- Group II (surgeon-only perioperative care program) (Active Comparator): Patients and their families meet with the surgeon at least once before surgery. After surgery, patients are managed daily during post-operative care. Patients may receive a referral for functional and nutritional prehabilitation at the discretion of the surgeon/surgical team. Patients and their families receive instructions to follow the standard procedures for reporting problems between clinic visits, including contacting their surgical team if symptoms become severe and physical function worsens; and the use of the hospital call line to report problems. Patients, caregivers and surgeons may receive the opportunity to participate in focus group in-person, via telephone, or videoconferencing.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Participate in a surgeon-only perioperative care program
  Other Names: standard of care; standard therapy
  Arms: Group II (surgeon-only perioperative care program)
Procedure: Functional Assessment — Complete a functional assessment
  Arms: Group I (telemonitoring program, actigraph, TapCloud)
Other: Medical Device Usage and Evaluation — Wear an actigraph
  Arms: Group I (telemonitoring program, actigraph, TapCloud)
Procedure: Nutritional Assessment — Complete a nutritional assessment
  Other Names: Dietary Assessment; dietary counseling; nutritional counseling
  Arms: Group I (telemonitoring program, actigraph, TapCloud)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: TapCloud — Use TapCloud app
  Arms: Group I (telemonitoring program, actigraph, TapCloud)

SUMMARY:
This phase III trial compares a home-based telemonitoring program that collects symptom and daily step information to surgeon only care in improving recovery and stopping complications within 30 days after surgery in patients with gastrointestinal, genitourinary, or gynecologic cancer who are scheduled to undergo abdominal surgery. Patients may experience a decrease in functional capacity and experience symptoms like pain and fatigue after surgery, and this may change their ability to walk and function. Home-based telemonitoring of patient symptoms and their ability to walk and function after surgery may help doctors and nurses find and treat problems early, which may improve the patient's recovery and lower the number of complications after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the impact of remote perioperative telemonitoring care versus surgeon only perioperative care on clinically significant changes in functional recovery (accelerometer daily step count) and related secondary patient-centered outcomes (sleep, sedentary time, symptom severity, symptom interference with daily activities).

II. Compare the impact of remote perioperative telemonitoring care versus surgeon only perioperative care on postoperative complications (Comprehensive Complications Index - CCI) and related secondary surgical outcomes (hospital readmission).

III. Compare early withdrawal (dropout or loss of accelerometer device) between the comparators.

IV. Explore perioperative telemonitoring care-related experiences (acceptability, technology usability, uptake/integration) among patients, families, and surgeons through qualitative focus groups and exit interviews.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (REMOTE PERIOPERATIVE TELEMONITORING CARE GROUP): Before surgery, patients complete a functional and nutritional assessment. The home environment of patients will also be assessed. Based on findings, patients undergo personalized prehabilitation. Patients also wear an actigraph throughout the study to measure and record daily steps taken and sedentary time. Patients use the TapCloud application (app) on a smart device (phone, tablet) or home computer to collect, track, and report their symptoms. Based on patient input in the TapCloud app, a real-time alert is sent to a registered nurse (RN) when predetermined thresholds are met. RNs then contact the patient via the TapCloud app and further phone calls if necessary. Patients, caregivers and surgeons may also participate in a focus group in-person, via telephone, or videoconferencing.

GROUP II (SURGEON ONLY PERIOPERATIVE CARE GROUP): Patients and their families meet with the surgeon at least once before surgery. After surgery, patients are managed daily during post-operative care. Patients may receive a referral for functional and nutritional prehabilitation at the discretion of the surgeon/surgical team. Patients and their families receive instructions to follow the standard procedures for reporting problems between clinic visits, including contacting their surgical team if symptoms become severe and physical function worsens; and the use of the hospital call line to report problems. Patients, caregivers and surgeons may receive the opportunity to participate in focus group in-person, via telephone, or videoconferencing.

After completion of study, patients are followed up for 3-4 months.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients scheduled to undergo major abdominal surgery for gastrointestinal (GI), genitourinary (GU), or gynecological (GYN) malignancies
* Ability to read and understand English or Spanish
* Patients across all stages of disease
* There are no restrictions related to performance status or life expectancy
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2026-11-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (3):
- United States (3):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope South Pasadena, South Pasadena, California

REFERENCES:
- [Derived] Sun V, Xiao Y, Li S, Palmer J, Tribby CP, Crane TE, Melstrom L, Dellinger T, Yuh B, Raz D, Cota-Robles E, Cota-Robles L, Nolde M, Ferrell B, Fong Y. Comparative effectiveness of remote perioperative telemonitoring in cancer surgery: a randomized trial. NPJ Digit Med. 2025 Aug 28;8(1):555. doi: 10.1038/s41746-025-01961-z. PMID 40877442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 398 participants were enrolled to the study, however 16 participants did not want to participate after signing consent and are considered attrition which is the reason why data analysis was done for 382 participants instead of the total consented/enrolled.
Pre-assignment Details: 398 participants were enrolled to the study, however 16 participants did not want to participate after signing consent and are considered attrition which is the reason why data analysis was done for 382 participants instead of the total consented/enrolled.
Period: Overall Study
Arm/Group | Group I (Telemonitoring Program, Actigraph, TapCloud) | Group II (Surgeon-only Perioperative Care Program)
Started | 189 | 193
Completed | 164 | 145
Not Completed | 25 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Telemonitoring Program, Actigraph, TapCloud) | Group II (Surgeon-only Perioperative Care Program) | Total
Number analyzed (Participants) | 189 | 193 | 382
Age, Continuous [Mean (Standard Deviation); unit: year] | 60.31 (11.72) | 60.90 (11.15) | 60.61 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 95 | 183
  Male | 101 | 98 | 199
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67 | 63 | 130
  Not Hispanic or Latino | 117 | 128 | 245
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 14 | 16 | 30
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 8 | 7 | 15
  White | 131 | 148 | 279
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 35 | 17 | 52
Region of Enrollment [Number; unit: participants]
  United States | 189 | 193 | 382

OUTCOME MEASURES:

1. Primary Outcome: Change in Daily Step Count
Description: Will calculate percent change from preoperative baseline in daily step count during the first 2 weeks post-discharge from hospital. Will use generalized linear mixed modeling (with treatment and covariates as fixed factors, patient identification as random factor).
Time Frame: Baseline up to day 14
Reporting Status: Not Posted, anticipated posting 2026-09

2. Primary Outcome: Time to Early Withdrawal
Description: Analyzed using proportional hazards regression.
Time Frame: Up to 4 months
Reporting Status: Not Posted, anticipated posting 2026-09

3. Primary Outcome: Qualitative Data
Description: Qualitative data from exit interviews and focus groups will be analyzed using the conventional content analysis approach.
Time Frame: Up to 4 months
Reporting Status: Not Posted

4. Primary Outcome: Post-operative Complications
Description: Assessed using the Comprehensive Complications Index (CCI) which summarizes the entire patient postoperative experience with respect to complications (on a scale from 0 to 100), and is based on the established Clavien-Dindo classification. For CCI score: Higher = worse
Time Frame: Up to 30 days after surgery
Population: 398 participants were enrolled to the study, however 16 participants did not want to participate after signing consent and are considered attrition which is the reason why data analysis was done for 382 participants instead of the total consented/enrolled. These number are accurate for analysis based on the data collection.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group I (Telemonitoring Program, Actigraph, TapCloud) | Group II (Surgeon-only Perioperative Care Program)
Number analyzed (Participants) | 189 | 193
units on a scale | 0 [0 to 42.4] | 0 [0 to 100]

5. Primary Outcome: Maximum CCI
Description: Maximum CCI will be categorized as above versus below 15, and logistic regression will be used to evaluate the effect of study intervention.
Time Frame: Up to 30 days post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Telemonitoring Program, Actigraph, TapCloud) | Group II (Surgeon-only Perioperative Care Program)
Number analyzed (Participants) | 189 | 193
Participants
  High (maximum CCI >= 15) | 14 | 20
  Low (maximum CCI < 15) | 167 | 155
  Missing due to attrition or no surgery scheduled | 8 | 18

6. Secondary Outcome: Time to Hospital Readmission
Description: Will be subjected to survival analysis.
Time Frame: Up to 90 days post-discharge
Reporting Status: Not Posted

7. Secondary Outcome: Change in Sedentary Time
Description: Assessed using the Actigraph GT9X Link. Data capture will focus on the following: 1) number of steps taken per day and 2) sedentary time. Recommended activity counts per minute (cpm) cutpoints will be used to categorize sedentary time (< 100 cpm) from light-intensity physical activity (100-1951 cpm) and moderate/vigorous intensity physical activity (>=1952 cpm).
Time Frame: Baseline up to 4 months
Reporting Status: Not Posted

8. Secondary Outcome: Change in General Symptoms
Description: Assessed using the MD Anderson Symptom Inventory.
Time Frame: Baseline up to 4 months
Reporting Status: Not Posted

9. Secondary Outcome: Change in Disease-specific Symptoms
Description: Assessed using the MD Anderson Symptom Library Items.
Time Frame: Baseline up to 4 months
Reporting Status: Not Posted

10. Secondary Outcome: Change in Sleep
Description: Assessed using the MD Anderson Symptom Inventory.
Time Frame: Baseline up to 4 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Since this is not a drug trial, there was no specific timepoint that was monitored for an adverse event to be recorded. It's an intervention trial that lasts 90 days post-treatment with no blood draws, procedures, etc. Patients were not assessed for specific adverse events however, 4 patients died during the study due to their ongoing cancer diagnosis, not due to study participation. The time frame where each participant was monitored/assessed for death was during the 90 days.
Description: Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed. Please see above regarding adverse events.
Arm/Group | Group I (Telemonitoring Program, Actigraph, TapCloud) | Group II (Surgeon-only Perioperative Care Program)
All-Cause Mortality (participants affected / at risk) | 0/189 | 4/193
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT04596384/Prot_SAP_000.pdf